CCF IRB #: 20-321 Approval Date: 4/10/2024 Expiration Date: 4/9/2025

### The Cleveland Clinic Foundation

# Consent to Participate in a Research Study

**Study title:** A Prospective Randomized Control Trial of The Effectiveness of Alvimopan as a Rescue Treatment of Postoperative Ileus Following Colorectal Surgery

Principal Investigator: Dr. Scott Steele (216-444-4715)

After hours phone contact #: During non-business hours call (216) 444-2200 and ask the operator to page the Colorectal Surgeon on call.

### **KEY INFORMATION**

The following is a short summary of this research study to help you decide whether or not to be a part of this research study. More detailed information is included later on in this document.

### What should I know about a research study?

- Someone will explain this research study to you.
- You can choose whether or not to take part.
- You can agree to take part and then later change your mind.
- Your decision whether or not to participate will not be held against you.
- You can ask all the questions you want before you decide.

## What is the purpose, procedures and duration of this study?

We invite you to take part in a research study because you have recently undergone surgery where part of your colon or small bowel was removed, or you had closure of your ileostomy, and now are experiencing a delay in regaining function of your gastrointestinal tract. The purpose of this study is to evaluate the effectiveness of the drug Alvimopan in the treatment of delayed return of gastrointestinal function.

Alvimopan is a drug that works by blocking receptors found in the gastrointestinal tract that can slow down the function of your gastrointestinal tract. It is approved by the Food and Drug Administration (FDA).

If you have been diagnosed with post-operative ileus, you will be randomized to receive the standard of care treatment or receive Alvimopan. If you are randomized to the Alvimopan group, you will be asked to ingest one to three Alvimopan tablets, 12 hours apart, and to answer questions about how you feel with regards to nausea, bloating, and about vomiting and bowel movements.

Your participation in the research will last about 30 days.

More detailed information can be found under the section labeled: "Information on the Research."

# Why might you choose not to participate in this research study?

You may not want to participate in this study if you have a history of indigestion, constipation, low blood levels of potassium, or low blood levels of iron.

More detailed information about the risks of this study can be found in the section labeled "Risks."

# Why might you choose to volunteer for this study?

We cannot know if you will have any benefit as a result of your participation in the study; it is possible the study treatment may improve your condition, which may give you relief from some symptoms or improve your quality of life. However, it is possible that your condition could worsen. Your participation in this study will help to obtain information about treating subjects with postoperative ileus (delayed return of gastrointestinal tract function after surgery).

More detailed information about the benefits of this study can be found in the section labeled "Benefits."

# What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example: The insertion of a nasogastric tube, which is a tube that is inserted through your nose into your stomach to allow the contents to be removed and to relieve bloating and nausea Not eating or drinking for a period of time until your symptoms improve

The alternative to being in this study is to not take part.

More detailed information about the alternatives to this study can be found in the section labeled "Alternatives."

#### **DETAILED INFORMATION**

The following is more detailed information about this study in addition to the information listed above.

### 1. INFORMATION ON THE RESEARCH

## Why is the research study being done?

Postoperative ileus, or delayed return of function of the gastrointestinal tract after surgery, is a common problem experienced by patients after surgery for removal of part of their colon or small bowel. Patients who experience this problem are more likely to have other medical problems during their hospitalization and are more likely to stay in the hospital for a longer period of time after surgery. Currently, there is no specific treatment for this condition. Studies have shown Alvimopan to be effective in treating this condition in some patients when given before and after surgery. It is possible that Alvimopan is more effective in patients who have already developed postoperative ileus. This study is being done to evaluate the effectiveness of Alvimopan in patients who are already experiencing a delayed return of gastrointestinal function after surgery.

Alvimopan was FDA approved in 2008 for short term use to speed up the return of gastrointestinal function after surgery where part of the colon or small bowel is removed.

## How Many People Will Take Part in this Study?

Approximately 58 people will take part in this study at Cleveland Clinic.

# What is involved if you decide to take part in this research study?

After your surgery you will be monitored for postoperative ileus (delayed return of function of your gastrointestinal tract). If you are diagnosed with postoperative ileus, you will be randomized to either the control group or the treatment group. Randomization is a process which will be used to assign you, by chance (like the flip of a coin), to one of the study groups. Neither you nor your doctor can choose which group you are in. Participants in the control group will receive standard of care for this condition and not the research treatment.

Participants in the treatment group will receive a maximum of 3 doses of Alvimopan 12mg orally, 12 hours apart. The first dose of Alvimopan will be given at the time of diagnosis of postoperative ileus, the second and/or third dose will only be given if symptoms do not resolve after the first dose. You will be continually monitored for symptoms such as nausea, vomiting, and bloating. Your ability to eat food and your bowel movements will also be recorded. The same criteria to determine when you are able to go home will be used for all participants in the study; you will be discharged home once you are deemed ready by your surgeon.

Your participation in this study will last about 30 days. Study information will be collected from your medical record and by direct contact with the health care providers taking care of you.

CCF IRB #: 20-321 Approval Date: 4/10/2024 Expiration Date: 4/9/2025

### How will my data be used?

The data we collect from you will be used to evaluate the effectiveness of Alvimopan in treating postoperative ileus compared to standard of care.

# 2. ALTERNATIVES

The alternative to being in this study is to not take part.

If you decide not to take part in this study, you have other choices. For example:

- The insertion of a nasogastric tube, which is a tube that is inserted through your nose into your stomach to allow the contents to be removed and to relieve bloating and nausea
- Not eating or drinking for a period of time until your symptoms improve

#### 3. RISKS

# What are the risks of participating in the research study?

Long-term use of Alvimopan is associated with an increased incidence of myocardial infarction (heart attack). Because of this, it is only approved for short-term use (15 doses), and in this study it will be used short-term for a maximum of 3 doses.

The most common side effect of Alvimopan is indigestion (1.5% of patients). Other side effects that you may experience include constipation, gas, low blood levels of potassium, low blood levels of iron, difficulty with urination, and back pain. The side effects caused by Alvimopan are mild in severity and temporary, and are readily treated in the hospital if required.

### Confidentiality Risks

There is a potential risk of loss of confidentiality of your data. Every effort will be made to keep your information confidential through the use of the following safeguards: data will be stored in a password protected computer accessible only by the research team, data will be collected in RedCap, a secure password protected data collection system. If you decide to be in this study, the study researchers will get information that identifies you and your personal health information. This may include information that might directly identify you, such as your name and address. This information will be kept for the length of the study. After that time it will be destroyed or de-identified, meaning we will replace your identifying information with a code that does not directly identify you. The principal investigator will keep a link that identifies you to your coded information, but this link will be kept secure and available only to the principal investigator or selected members of the research team. Any information that can identify you will remain confidential. Any personal information that could identify you will be removed or changed before files are shared with other researchers or results are made public.

#### 4. BENEFITS

Participation in this study may help to improve your condition, but it is also possible that your condition may worsen. There is no guarantee that you will personally benefit by participating in this research study. Your participation in this study may provide information that may help other people who have a similar medical problem in the future.

#### 5. COSTS

There is no cost to you to be in this research study.

#### 6. PAYMENT

You will not receive any payment if you participate in this study.

#### 7. RESEARCH RELATED INJURY

There is minimal risk to you if you take part in this research.

#### 8. PRIVACY AND CONFIDENTIALITY

## What will happen to your information that is collected for this research?

Cleveland Clinic may share your study information, without anyone knowing that it is related to you specifically, with others or use it to research projects not listed in this form. Your data may be stored and shared for future research without additional informed consent if identifiable private information, such as your name and medical record number, are removed. If your identifying information is removed from your data, we will no longer be able to identify and destroy them.

Study results may be shared in medical journals, at scientific meetings, and in other mediums without your identifying information. Your records will be confidential and your identity will not be shared in medical journals, at scientific meetings, and in other mediums without your express consent.

### Authorization to Use/Disclose Protected Health Information

Cleveland Clinic has rules and procedures to protect information about you. Federal and State laws also protect your privacy.

The research team working on the study will collect information about you. This includes your health information, data collected for this research study and personal identifying information including your name, address, date of birth and other identifying information.

Generally, only people on the research team will know your identity and that you are in the research study. However, sometimes other people at Cleveland Clinic may see or give out your

information. These include people who review research studies including the Institutional Review Board and Research Compliance, their staff, lawyers, or other Cleveland Clinic staff.

People outside Cleveland Clinic may see your information for this study. Examples include government groups (such as the Food and Drug Administration), safety monitors, other hospitals in the study and the sponsor of the research and their agents. Cleveland Clinic will do our best to ensure your information is kept confidential and that only the health information which is minimally required to conduct the study is used or disclosed to people outside Cleveland Clinic; however, people outside Cleveland Clinic who receive your information may not be covered by this promise.

You do not have to give this permission to use and give out your information; however you will not be able to participate in this research study without providing this permission by signing this consent form. The use and disclosure of your information has no expiration date.

You may cancel your permission to use and disclose your information at any time by notifying the Principal Investigator in writing, Dr. Scott Steele at Crile Building, A-100, 2049 East 100<sup>th</sup> Street, Cleveland, OH, 44195. If you do cancel your permission to use and disclose your information, your participation in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in the study.

#### Clinical Trials Language

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U. S. law. This Website will not include information that can identify you. At most, the Website will include a summary of the results. You can search the Website at any time.

# 9. QUESTIONS

If you have any questions or concerns about the research, or develop a research-related problem, you should contact Dr. Scott Steele at 216-444-4715, Crile Building, A-100, 2049 East 100<sup>th</sup> Street, Cleveland, OH, 44195. During non-business hours, weekends and holidays, please call (216) 444-2200 and ask the operator to page the Colorectal Surgeon on call. If you have questions about your rights as a research subject, you should contact the Institutional Review Board at (216) 444-2924.

#### 10. VOLUNTARY PARTICIPATION

### What are your rights as a research participant?

Taking part in this study is voluntary. You will be told of any new, relevant information from the research that may affect your health, welfare, or willingness to continue in this study. You may choose not to take part or may leave the study at any time. Withdrawing from the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to withdraw from the study you should discuss with your study doctor your decision to ensure a safe withdrawal.

CCF IRB #: 20-321 Approval Date: 4/10/2024 Expiration Date: 4/9/2025

If you leave the study early, Cleveland Clinic may use or give out your health information that it has already collected if the information is needed for this study or any follow-up activities.

Your refusal to participate will not prejudice your future treatment or benefits here at the Cleveland Clinic. You may discontinue participation in the study at any time without fear of penalty or loss of medical care. If you decide to withdraw from the study you can contact the principal investigator of this study, Dr. Scott Steele at 216-444-4715, Crile Building, A-100, 2049 East 100<sup>th</sup> Street, Cleveland, OH, 44195

### Subject's Withdrawal from the Study

You may withdraw from this study at any time during your hospitalization or after discharge from the hospital.

#### 11. SIGNATURES

Statement of Participant

I have read and have had verbally explained to me the above information and have had all my questions answered to my satisfaction. I understand that my participation is voluntary and that I may stop my participation in the study at any time. Signing this form does not waive any of my legal rights. I understand that a copy of this consent will be provided to me. By signing below, I agree to take part in this research study.

| Printed name of Participant | | | |
|---|---|---|---|
| Participant Signature | Date | s | |
| Statement of Person Conducting Info | rmed Consent Dis | cussion | |
| I have discussed the information contain opinion that the participant understands with this research study. | | | ed |
| Printed name of person obtaining conser | nt | | |
| Signature of person obtaining consent | Date | e | |

......

\_\_\_\_\_